CLINICAL TRIAL: NCT05473013
Title: Optimizing Digital Health Technologies to Improve Therapeutic Skill Use and Acquisition
Brief Title: Optimizing Digital Health Technology Interventions to Increase Skill Acquisition and Utilization
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Drexel University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 2201009012; R01MH129478 (NIH)
Record Dates: First submitted 2022-07-18; First posted 2022-07-25 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: Bulimia Nervosa; Bulimia; Binge Eating; Binge-Eating Disorder
Keywords: Eating disorders; Bulimia Nervosa; Bulimia; Binge Eating; Binge Eating Disorder; Cognitive Behavioral Treatment for Eating Disorders; Digital health technologies (DHTs); Micro-Interventions
MeSH Terms: conditions — Bulimia Nervosa; Bulimia; Binge-Eating Disorder; Feeding and Eating Disorders | interventions — Behavior Therapy

STUDY DESIGN:
Intervention Model Description: MOST: multiphase optimization strategy
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Base BT (Skills Monitoring Off + No Micro-Interventions) (Active Comparator): 16 weekly sessions of standard behavioral therapy for eating disorders aimed at changing behaviors that maintain binge eating (e.g. rigid dietary restriction outside of binge episodes, irregular or chaotic eating patterns). This will include traditional self-monitoring of participants' eating patterns, binging, and (if applicable) compensatory behaviors via a smartphone application.
  Interventions: Behavioral: Behavioral Therapy for Eating Disorders
- Base BT + Skills Monitoring On + No Micro-Interventions (Experimental): 16 weekly sessions of standard behavioral therapy for eating disorders aimed at changing behaviors that maintain binge eating (e.g. rigid dietary restriction outside of binge episodes, irregular or chaotic eating patterns). This will include a more complex self-monitoring than the self-monitoring protocol with traditional behavioral treatment. Via a smartphone application, participants will be asked to self-monitor skill usage of the skills provided during treatment sessions on top of monitoring their eating patterns, binging, and (if applicable) compensatory behaviors.
  Interventions: Behavioral: Behavioral Therapy for Eating Disorders; Behavioral: Skills Monitoring On
- Base BT + Skills Monitoring On + Automated Reminder Messages (Experimental): 16 weekly sessions of standard behavioral therapy for eating disorders aimed at changing behaviors that maintain binge eating (e.g. rigid dietary restriction outside of binge episodes, irregular or chaotic eating patterns).This will include a more complex self-monitoring than the self-monitoring protocol with traditional behavioral treatment. Via a smartphone application, participants will be asked to self-monitor skill usage of the skills provided during treatment sessions on top of monitoring their eating patterns, binging, and (if applicable) compensatory behaviors. It will also include participants receiving two randomly time automated push notifications from the application each week to remind them about skills they have learned in session to encourage skill use.
  Interventions: Behavioral: Behavioral Therapy for Eating Disorders; Behavioral: Skills Monitoring On; Behavioral: Automated Reminder Messages
- Base BT + Skills Monitoring On + JITAIs (Experimental): 16 weekly sessions of standard behavioral therapy for eating disorders aimed at changing behaviors that maintain binge eating (e.g. rigid dietary restriction outside of binge episodes, irregular or chaotic eating patterns). This will include a more complex self-monitoring than the self-monitoring protocol with traditional behavioral treatment. Via a smartphone application, participants will be asked to self-monitor skill usage of the skills provided during treatment sessions on top of monitoring their eating patterns, binging, and (if applicable) compensatory behaviors. It will also include participants receiving push notifications each week to remind them about skills they have learned in session to encourage skill use during app-identified moments of need (i.e., JITAIs, just-in-time adaptive interventions).
  Interventions: Behavioral: Behavioral Therapy for Eating Disorders; Behavioral: Skills Monitoring On; Behavioral: JITAIs
- Base BT + Skills Monitoring Off + Automated Reminder Messages (Experimental): 16 weekly sessions of standard behavioral therapy for eating disorders aimed at changing behaviors that maintain binge eating (e.g. rigid dietary restriction outside of binge episodes, irregular or chaotic eating patterns). This will include traditional self-monitoring of participants' eating patterns, binging, and (if applicable) compensatory behaviors via a smartphone application. It will also include participants receiving two randomly time automated push notifications from the application each week to remind them about skills they have learned in session to encourage skill use.
  Interventions: Behavioral: Behavioral Therapy for Eating Disorders; Behavioral: Automated Reminder Messages
- Base BT + Skills Monitoring Off + JITAIs (Experimental): 16 weekly sessions of standard behavioral therapy for eating disorders aimed at changing behaviors that maintain binge eating (e.g. rigid dietary restriction outside of binge episodes, irregular or chaotic eating patterns). This will include traditional self-monitoring of participants' eating patterns, binging, and (if applicable) compensatory behaviors via a smartphone application. It will also include participants receiving push notifications each week to remind them about skills they have learned in session to encourage skill use during app-identified moments of need (i.e., JITAIs, just-in-time adaptive interventions).
  Interventions: Behavioral: Behavioral Therapy for Eating Disorders; Behavioral: JITAIs

INTERVENTIONS:
Behavioral: Behavioral Therapy for Eating Disorders — Standard behavioral therapy for eating disorders aimed at changing behaviors that maintain binge eating (e.g. rigid dietary restriction outside of binge episodes, irregular or chaotic eating patterns).
Behavioral: Skills Monitoring On — Integrates behavioral treatment for eating disorders with a more complex self-monitoring than the self-monitoring protocol with traditional behavioral treatment. Via a smartphone application, participants will be asked to self-monitor skill usage of the skills provided during treatment sessions on top of monitoring their eating patterns, binging, and (if applicable) compensatory behaviors.
  Other Names: Enhanced Skills Monitoring
  Arms: Base BT + Skills Monitoring On + Automated Reminder Messages; Base BT + Skills Monitoring On + JITAIs; Base BT + Skills Monitoring On + No Micro-Interventions
Behavioral: Automated Reminder Messages — Integrates behavioral treatment for eating disorders with two randomly time automated push notifications from a smartphone application each week to remind participants about skills they have learned in session to encourage skill use.
  Other Names: Micro-Intervention 1
  Arms: Base BT + Skills Monitoring Off + Automated Reminder Messages; Base BT + Skills Monitoring On + Automated Reminder Messages
Behavioral: JITAIs — Integrates behavioral treatment for eating disorders with push notifications each week from a smartphone application to remind participants about skills they have learned in session to encourage skill use during app-identified moments of need (i.e., JITAIs, just-in-time adaptive interventions).
  Other Names: Micro-Intervention 2
  Arms: Base BT + Skills Monitoring Off + JITAIs; Base BT + Skills Monitoring On + JITAIs

SUMMARY:
The purpose of this study is to identify the independent and combined effects of two types of self-monitoring and two types of micro-interventions when combined with standard cognitive behavioral treatment for bulimia nervosa (BN) and binge eating disorder (BED). The primary aims of this study are (1) to evaluate the optimal complexity of Self-Monitoring and Micro-Interventions on eating pathology (at post-treatment and at 6 and 12-month follow-ups and (2) to test the hypotheses that the optimal complexity level of each component is moderated by baseline deficits in self-regulation. The secondary aim will be to test target engagement for each level of complexity for each component, i.e., to test whether higher complexity of each technological components is associated with better rates of therapeutic skill use and acquisition and that improvements in skill use and acquisition are associated with improvements in outcomes. A final exploratory aim will be to quantify the component interaction effects, which may be partially additive (because components overlap and/or there is diminishing return), fully additive, or synergistic (in that component complexities may partially depend on each other).

DETAILED DESCRIPTION:
The current study will use a 2 x 3 full factorial design in which 264 individuals with BN or BED are assigned to one of six treatment conditions, i.e., representing each permutation of self-monitoring complexity (Skills-Monitoring On vs. Skills-Monitoring Off) and micro-intervention complexity (No Micro-Interventions vs. Automated Reminder Messages vs. JITAIs) as an augmentation to CBT. All participants will be given the gold-standard treatment for eating disorders known as cognitive behavioral therapy (CBT-E) which is the most evidence-based treatment to date for eating disorders and is a well-established treatment approach. The main innovation of the new proposed study is the evaluation of the efficacy of the six intervention conditions that arise as a result of testing each possible combination of self-monitoring complexity (Skills-Monitoring On vs. Skills-Monitoring Off) and micro-intervention complexity (No Micro-Interventions vs. Automated Reminder Messages vs. JITAIs) as an augmentation to CBT.

The purpose of this study is to identify the independent and combined effects of two types of self-monitoring and two types of micro-interventions when combined with standard cognitive behavioral treatment for bulimia nervosa (BN) and binge eating disorder (BED). The primary aims of this study are (1) to evaluate the optimal complexity of Self-Monitoring and Micro-Interventions on eating pathology (at post-treatment and at 6 and 12-month follow-ups and (2) to test the hypotheses that the optimal complexity level of each component is moderated by baseline deficits in self-regulation. The secondary aim will be to test target engagement for each level of complexity for each component, i.e., to test whether higher complexity of each technological components is associated with better rates of therapeutic skill use and acquisition and that improvements in skill use and acquisition are associated with improvements in outcomes. A final exploratory aim will be to quantify the component interaction effects, which may be partially additive (because components overlap and/or there is diminishing return), fully additive, or synergistic (in that component complexities may partially depend on each other).

ELIGIBILITY:
Inclusion Criteria:

1. Have experienced 12 or more loss of control episodes within the previous 3 months
2. Have a BMI at or above 18.5
3. Are located in the US and willing/able to participate in treatment and assessments
4. Are able to give consent

Exclusion Criteria:

1. Are unable to fluently speak, write and read English
2. Have a BMI below 18.5
3. Are already receiving treatment for an eating disorder
4. Require immediate treatment for medical complications as a result of eating disorder symptoms
5. Have a mental handicap, or are experiencing other severe psychopathology that would limit the participants' ability to comply with the demands of the current study (e.g. severe depression with suicidal intent, active psychotic disorder, severe substance use)
6. Are pregnant or are planning to become pregnant

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Estimated)
Dates: Start 2023-01-06 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Binge eating frequency assessed by the Eating Disorder Examination | Changes from each assessment time point throughout treatment (3 assessments over 16 weeks) and at a 6 month and a 12-month post-treatment follow-up assessment
  Frequency (number of days and number of instances) of binge eating over the past 28 days assessed by the Eating Disorder Examination
Global Eating Pathology | Changes from each assessment time point throughout treatment (3 assessments over 16 weeks) and at a 6 month and a 12-month post-treatment follow-up assessment
  The Eating Disorder Examination is a semi-structured interview that measures eating. pathology. The EDE yields a total eating pathology score that will be used as an outcome variable. Global eating pathology is on a 0-6 point scale with higher scores indicating more significant eating pathology.
Remission Status | Changes from each assessment time point throughout treatment (3 assessments over 16 weeks) and at a 6 month and a 12-month post-treatment follow-up assessment
  Presence or absence of eating disorder diagnosis. Not in remission; in partial remission; or in full remission.
BMI | Changes from each assessment time point throughout treatment (3 assessments over 16 weeks) and at a 6 month and a 12-month post-treatment follow-up assessment
  kilogram/(meters^2), this will be calculated by assessors when participants provide their height and weight at all assessment points

SECONDARY OUTCOMES:
Compensatory behavior frequency assessed by the Eating Disorder Examination (EDE) | Changes from each assessment time point throughout treatment (3 assessments over 16 weeks) and at a 6 month and a 12-month post-treatment follow-up assessment
  Frequency (number of days and number of instances) of compensatory behaviors assessed by the Eating Disorder Examination
Acceptability and Feasibility | Changes from each assessment time point throughout treatment after baseline so 2 assessments over 16 weeks (the mid-treatment and post-treatment assessments).
  Perceived usefulness and ease-of-use of the technological components (the smartphone application) will be measured by the Technology Acceptance Model (TAM) Scales. A Feedback Questionnaire will also be used to measure qualitative acceptability of both the technological components of the study and the treatment components. Assessment of feasibility will include % of eligible patients enrolled, treatment attrition (% of patients that prematurely terminate treatment), and study retention (% of patients that complete all assessment points). Data will also be collected on participants' use of CBT+ technological features, including time, duration, and frequency of use.
Frequency of skill use and success of skill use | Changes from each weekly session over the course of the 16 week treatment
  Data will be collected at each therapy session via a pre-session questionnaire for participants and post-session questionnaire for therapists to assess skills related to internal experiences such as urges and negative emotions that contribute to ED behaviors. The items were adapted from the Difficulties in Emotional Regulation Scale (DERS).
Emotional Self-regulation | Changes from each assessment time point throughout treatment (3 assessments over 16 weeks) and at a 6 month and a 12-month post-treatment follow-up assessment
  Changes in emotional self-regulation will be assessed using the total score of the Difficulties in Emotional Regulation Scale (DERS)
Self-regulation: Impulsivity | Changes from each assessment time point throughout treatment (3 assessments over 16 weeks) and at a 6 month and a 12-month post-treatment follow-up assessment
  Changes in impulsivity will be assessed by the total score of the UPPS-P Impulsive Behaviors Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Adrienne S Juarascio, Ph.D., Principal Investigator — Drexel University
Locations (1):
- Drexel University, Stratton Hall, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
We will follow all guidelines for data sharing through the National Database for Clinical Trials Related to Mental Illness (NDCT) and the NIMH Data Archive (NDA). All de-identified data will be submitted to the NDA at the item level and subject level.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Within one year of project completion
Access Criteria: We will include supporting documentation to allow other researchers to use this data easily and appropriately.

REFERENCES:
- [Derived] Juarascio AS, Presseller EK, Trainor C, Boda S, Manasse SM, Srivastava P, Forman EM, Zhang F. Optimizing digital health technologies to improve therapeutic skill use and acquisition alongside enhanced cognitive-behavior therapy for binge-spectrum eating disorders: Protocol for a randomized controlled trial. Int J Eat Disord. 2023 Feb;56(2):470-477. doi: 10.1002/eat.23864. Epub 2022 Nov 30. PMID 36448475